CLINICAL TRIAL: NCT02326766
Title: Blood Pressure Lowering Effect of Supplementation With Korea Red Ginseng Associated With Reductions in Circulating Lp-PLA2 Activity and Lysophospatidylcholines and an Increase in Dihydrobiopterin in Prehypertensive Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KGC_metabolites_14121
Record Dates: First submitted 2014-12-22; First posted 2014-12-29 (Estimated); Last update posted 2014-12-29 (Estimated); Status verified 2014-12

CONDITIONS: Prehypertension
MeSH Terms: conditions — Prehypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- KRG (Experimental): 5g Korea red ginseng (KRG)
  Interventions: Dietary Supplement: KRG
- Placebo (Placebo Comparator): 5 g placebo (corn starch)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: KRG — 5g Korea red ginseng (KRG)
  Arms: KRG
Dietary Supplement: Placebo — 5g placebo
  Arms: Placebo

SUMMARY:
This study evaluated effects of red ginseng consumption on blood pressure (BP) and fasting plasma metabolomes.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled study was conducted on nonobese, nondiabetic and prehypertensive subjects. Over a 12 week test period, the red ginseng group (n=31) consumed 10 capsules (total 5g) daily containing red ginseng, while the placebo group (n=31) consumed the same product without red ginseng. Fasting plasma metabolomes were profiled using UPLC-LTQ-Orbitrap mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* nondiabetic, nonobese and prehypertensive subjects with blood pressures ranging 120 - 139 mmHg (systolic) or 80-89 mmHg (diastolic) were enrolled in this study.

Exclusion Criteria:

* exclusion criteria included previous diagnosed clinical hypertension
* self-reported use of antihypertensive medication
* abnormal liver or renal function
* history of cardiovascular disease
* kidney disease
* cancer
* thyroid or pituitary disease or any other serious life-threatening illness that required regular medical treatment
* we also excluded women who were pregnant, breast feeding or intending to become pregnant during the time of study.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2011-11; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
changes from baselilne in blood pressure | 12 week

SECONDARY OUTCOMES:
changes from baseline in plasma metabolites | 12 week

REFERENCES:
- [Derived] Cha TW, Kim M, Kim M, Chae JS, Lee JH. Blood pressure-lowering effect of Korean red ginseng associated with decreased circulating Lp-PLA2 activity and lysophosphatidylcholines and increased dihydrobiopterin level in prehypertensive subjects. Hypertens Res. 2016 Jun;39(6):449-56. doi: 10.1038/hr.2016.7. Epub 2016 Feb 4. PMID 26843120